CLINICAL TRIAL: NCT04622020
Title: Effectiveness of Ultrasound Guided Intermediate Cervical Plexus Block (iCPB) in Patients With Refractory Chronic Neck Pain From Whiplash Associated Disorder (WAD): an Observational Study
Brief Title: Cervical Plexus Block (CPB) in Whiplash Associated Disorder (WAD)
Status: Completed | Type: Observational
Sponsor: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: EDGE 129250
Record Dates: First submitted 2020-11-01; First posted 2020-11-09 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2022-05

CONDITIONS: Whiplash Associated Disorder
Keywords: Cervical Plexus Block; Whiplash injury; WAD
MeSH Terms: conditions — Whiplash Injuries | interventions — Cervical Plexus Block; Anesthesia, Local

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients with chronic neck pain (> 3 months) following whiplash injury: Cervical plexus block with local anaesthesia followed by Cervical Plexus block with depot steroids
  Interventions: Procedure: Cervical Plexus Block with Local Anaesthesia; Procedure: Cervical Plexus Block with Depot Steroids

INTERVENTIONS:
Procedure: Cervical Plexus Block with Local Anaesthesia — Ultrasound guided intermediate cervical plexus block
Procedure: Cervical Plexus Block with Depot Steroids — Ultrasound guided intermediate cervical plexus block

SUMMARY:
Whiplash is the most common injury associated with motor vehicle accidents and a major cause of disability and litigation. An acute whiplash injury follows sudden or excessive hyperextension, hyper flexion, or rotation of the neck affecting the soft tissues. It typically results from rear-end or side-impact motor vehicle collisions. Patients commonly present with pain and stiffness in the neck, headache, and upper backache. Chronic whiplash syndrome is characterized by symptoms of neck pain that persist for more than 3 months (1, 2). With over half a million people making whiplash injury claims per annum in the UK, it has a major impact on the healthcare and legal systems and also the economy. Over 40% of patients with whiplash injury report chronic neck pain and this is often refractory to conservative management (pain relief medications, physiotherapy). Current treatment involves burning the small nerves that supply the joints (facet joints) in the neck. Although they provide pain relief that can last 6-9 months, the nerves re-grow and the treatment has to be repeated. This treatment is a complex procedure that requires extensive training and has the potential to cause serious harm. There is new evidence to show that the pain in whiplash injury could be due to an impaired function of the neck muscles arising from whiplash trauma. Current treatment for this condition is injection of numbing medicine or steroids directly into the muscle. Although this treatment is safer than burning the facet nerves, it provides short-term relief.

The investigators have shown that a novel treatment targeting the nerves that supply the muscles in the neck can provide durable relief in patients with chronic neck pain. The medication is injected into a specific area (plane) in the neck of the patient and is called cervical plexus block (CPB). The investigators currently offer CBP treatment as a standard treatment in the management of patients with chronic neck pain arising from whiplash injury. There are two types of CPB: CPB with numbing medicine (CPB-LA) and CPB with steroid.

Aim of the study is to evaluate the effectiveness of two types of Cervical Plexus Block (CPB) treatment in reducing pain at three months in patients with refractory chronic neck pain from whiplash injury

Methods: The proposed study is a prospective, observational pilot study that will be conducted at Leicester General Hospital over 36 months. Potential participants will be given an information sheet by the clinical team when they are seen in the outpatient clinic. The participants will have 24 hours to read the information sheet. Thereafter, the research team will approach the potential participant to obtain informed consent. After providing written consent, adult patients with chronic neck pain from whiplash injury will receive ultrasound guided CPB-LA in the theatre. If treatment provides >30% relief at 3 months, they will be re-assessed at six months and CPB-LAi will be repeated as per waiting list. If at 3 months, the pain returns to the baseline, CPB with steroid will be performed. If CPB with steroid does not provide any benefit, the participants will receive a rescue treatment (trigger point injection) within three months. Participants will be asked to complete questionnaires on pain scores and mood. Participation in the study will end at 9 months following the first CPB treatment on completion of relevant questionnaires.

DETAILED DESCRIPTION:
Whiplash is the most common injury associated with motor vehicle accidents and a major cause of disability and litigation. An acute whiplash injury follows sudden or excessive hyperextension, hyper flexion, or rotation of the neck affecting the soft tissues. It typically results from rear-end or side-impact motor vehicle collisions. Patients commonly present with pain and stiffness in the neck, headache, and upper backache with or without paraesthesia of the upper limbs. Chronic whiplash syndrome is characterized by symptoms that persist for more than 3 months. With over half a million people making whiplash injury claims per annum in the UK, it has a major impact on the healthcare and legal systems and also the economy. In 1995, whiplash-associated disorder (WAD) was defined by the Quebec task force as 'Whiplash is an acceleration-deceleration mechanism of energy transfer to the neck. The incidence of WAD is very variable, averaging to about 9 per 1000 people in the UK, the highest in Europe.

Around 40% of patients suffer from symptoms of WAD beyond 3 months (chronic whiplash) and 2 - 4.5% of patients are left permanently disabled.

There is evidence that neck pain in WAD could arise from either cervical facet joint or due to impaired function of neck muscles (Cervicothoracic Myofascial Pain Syndrome, CTMPS) or both. The investigators have recently reported on ultrasound guided cervical plexus block with depot steroids in the management of refractory cervicothoracic myofascial pain. This intervention involves a single injection that targets a number of muscles that are commonly involved in causing chronic WAD. The treatment has a definite end point that helps to standardize the intervention with a good safety profile.

The present study is an observational study on the effectiveness of two types of cervical plexus block (CPB-Local Anaesthesia and CPB-Steroids) treatment as a part of standard care in providing durable analgesia. The objective is to collect data to inform the design a larger multicentre study

ELIGIBILITY:
Inclusion Criteria:

1. All patients aged over 18 years and under 90 years willing to consent
2. History of whiplash injury
3. Chronic neck pain for above 3 months
4. Moderate to severe pain in the neck: Baseline NRS >4 (worst pain the last 24 hours)

Exclusion Criteria:

1. Lack of consent, including from those patients who lack mental capacity to give informed consent.
2. Past History of chronic neck pain that was present before suffering a whiplash injury
3. Patients with known history of drug allergy to depomedrone
4. Patients with infection at injection site at on day of treatment
5. Patients aged under 18 years or over 90 years
6. Unwilling to provide consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is based on a cohort of adult patients present with chronic neck pain arising from whiplash injury Chronic Neck Pain is defined as persistent neck pain that lasts for more than three months.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-06-26 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2022-08-20 (Actual)

PRIMARY OUTCOMES:
Primary outcome will be Pain at its Worst in the last 24 hours at the baseline and 3 months following the interventional treatment | 3 months
  Effective outcome: A two-point change in the Numerical Rating Scale (Pain at its worst in the last 24 hours) at three months when compared to the baseline. The Pain at its worst in 24 hours will be measured on the Brief Pain Inventory-short form (BPI-SF) question number 3 on Brief Pain Inventory -short form questionnaire. The expected change is a

SECONDARY OUTCOMES:
Treatment Failure rate: absence of sustained benefit at three month follow up | 3 months
  No reduction in NRS 'Pain at its worst in the last 24 hours' at three months when compared to the baseline NRS
Pain at its Worst in the last 24 hours at the baseline and 6 months | 6 months
  Change in the Pain at its worst score at 6 months when compared to the baseline
Change in Neck Disability Index (NDI) at 3 and 6 months when compared to baseline | 6 months
  Change in neck disability index at three and 6 months when compared to the baseline scoree that is measured on the NDI questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: G Niraj, MD, Principal Investigator — University Hospitals, Leicester
Locations (1):
- University Hospitals of Leicester NHS Trust, Leicester, United Kingdom